CLINICAL TRIAL: NCT00981110
Title: Surgical Sites Infections Following Colorectal Cancer Surgery. A Randomized Prospective Trial Comparing Standard and Advanced Antimicrobial Dressing Containing Ionic Silver.
Brief Title: Standard Versus Advanced Antimicrobial Dressing Containing Ionic Silver Following Colorectal Cancer Surgery
Acronym: AM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IEO S402/208
Record Dates: First submitted 2009-08-31; First posted 2009-09-22 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Colorectal Cancer
Keywords: Surgical site infections (SSI); Advanced antimicrobial dressing and clean surgery; Hydrofibre dressing
MeSH Terms: conditions — Colorectal Neoplasms; Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mepore Self-adhesive absorbent dressing (Active Comparator): Mepore Self-adhesive absorbent dressing
  Interventions: Device: Mepore Self-adhesive absorbent dressing
- AQUAGEL Ag Hydrofiber Wound Dressing (Experimental): AQUAGEL Ag Hydrofiber Wound Dressing
  Interventions: Device: AQUAGEL Ag Hydrofiber Wound Dressing

INTERVENTIONS:
Device: AQUAGEL Ag Hydrofiber Wound Dressing — Hydrofibre dressing containing ionic silver: medication performed as for frequency and duration according standard procedure
  Other Names: AQUAGEL Ag Hydrofiber Wound Dressing (ConvaTee,US)
  Arms: AQUAGEL Ag Hydrofiber Wound Dressing
Device: Mepore Self-adhesive absorbent dressing — Standard dressing: medication performed as for frequency and duration according standard procedure
  Arms: Mepore Self-adhesive absorbent dressing

SUMMARY:
The purpose of this study is to evaluate the efficacy of treatment with hydrofibre dressing in comparison with the efficacy of standard dressing in terms of prevalence of surgical site infections (SSI) in patients who underwent colorectal resection for malignancy.

ELIGIBILITY:
Inclusion Criteria:

* Patients bearing solid tumours who are candidate to open radical surgery for colorectal cancer (histology proven)
* Age 18-75
* Informed signed consent
* Performance Status 0-2 (according to ECOG score)
* Platelets > 50.000/mm3
* Prothrombin Time (Quick) > 60%
* White Blood Cells > 2500/mm3
* Life Expectancy > 3 months

Exclusion Criteria:

* Intestinal obstruction
* Severe intestinal bleeding requiring blood transfusion
* Age under 18 or over 75
* Severe hepatic failure (ascites, portal hypertension, jaundice or encephalopathy)
* Renal failure (hemodialysis, creatinin > 2.5 mg/dL)
* Active infections
* Coagulopathy
* Inability to give an informed consent
* Known allergies to dressing components

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-06; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The rate of patients with a Surgical site infection | 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Andreoni, MD, Principal Investigator — European Institute of Oncology; Roberto Biffi, MD, Principal Investigator — European Institute of Oncology; Emilio Bertani, MD, Principal Investigator — European Institute of Oncolgy
Locations (2):
- Italy (2):
  - S. Gerardo Hospital, Monza, Monza
  - European Institute of Oncology, Milan

REFERENCES:
- [Derived] Biffi R, Fattori L, Bertani E, Radice D, Rotmensz N, Misitano P, Cenciarelli S, Chiappa A, Tadini L, Mancini M, Pesenti G, Andreoni B, Nespoli A. Surgical site infections following colorectal cancer surgery: a randomized prospective trial comparing common and advanced antimicrobial dressing containing ionic silver. World J Surg Oncol. 2012 May 23;10:94. doi: 10.1186/1477-7819-10-94. PMID 22621779